CLINICAL TRIAL: NCT06634355
Title: Placental Transfer of Sugammadex in the Human Placental Perfusion Model
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S54819(ML8732)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy
Keywords: sugammadex; ex-vivo placenta perfusion model; placental transfer; pregnancy; anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ex-vivo placenta perfusion (Experimental): Measurement of placental transfer.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — In an ex-vivo placenta perfusion study, placental transfer of sugammadex is measured.

SUMMARY:
Preclinical research raised concern regarding the foetal effects of using sugammadex during pregnancy. However, to the best of our knowledge, the placental transfer of sugammadex has never been measured. As these data would be critical in assessing the foetal effects after maternal administration of sugammadex, it is warranted to measure the placental transfer of sugammadex. The aim of this project is to measure the placental transfer of sugammadex in the human placenta by using the ex vivo human placenta perfusion model.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed
* (placenta of a) pregnant women with an uncomplicated pregnancy and delivery

Exclusion Criteria:

* chronic medication use during pregnancy
* maternal diseases during pregnancy (including diabetes mellitus, hypertension, thyroid dysfunction), or any infection (chorioamnionitis and toxoplasmosis, other, rubella, cytomegalovirus, herpes infections, or a positive anti-HIV, anti-hepatitis B virus, or anti-hepatitis C virus serology)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Foetal-maternal ratio of the drug | On the same day as collection of placenta
  Drug concentrations of samples from the maternal and fetal compartment in the ex-vivo placenta perfusion model will be determined by high performance liquid chromatography and mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Kristel Van Calsteren, MD, PhD, Principal Investigator — University Hospital, Gasthuisberg; Sarah Devroe, MD, Phd, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No